CLINICAL TRIAL: NCT00664989
Title: Resurfacing Hemiarthroplasty Versus Conventional Stemmed Hemiarthroplasty
Brief Title: Resurfacing Hemiarthoplasty Versus Conventional Stemmed Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: 2006867-01H
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
Keywords: Hemiarthroplasty Stemmed Resurfacing Conventional Shoulder
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis: What is the difference in disease specific quality of life between patients who receive a humeral surface replacement hemiarthroplasty verusu a conventioanl stemmed hemiarthroplasty

DETAILED DESCRIPTION:
The purpose of this multi-centered, randomized, controlled trial will be to determine if patient self-assessed outcomes (Western Ontario Osteoarthritis of Shoulder Score- WOOS) following humeral resurfacing are superior to those following a conventional, modular, stemmed, humeral prosthesis. The first phase of this study will be a one year pilot recruitment period. This is necessary in order to determine both a center by center, and national recruitment rate, and to determine a sample size necessary for a sufficiently powered full randomized trial. If a full randomized trial is not considered feasible following Phase 1, then a prospective cohort study will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Recent humeral resurfacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: recent humeral resurfacing
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — OHRI
Locations (1):
- OHRI, Ottawa, Ontario, Canada